CLINICAL TRIAL: NCT00752115
Title: Randomized Phase II Study of Combination Chemotherapy With Sildenafil Plus Carboplatin and Weekly Paclitaxel in Patients With Previously Untreated Advanced Non-small Cell Lung Cancer
Brief Title: Combination Chemotherapy With Sildenafil Plus Carboplatin and Paclitaxel in Patients With Advanced Non-small Cell Lung Cancer
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Hamamatsu University (Other)
Responsible Party: Principal Investigator, Naoki Inui, Department of Respiratory Medicine, Hamamatsu University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Hamamatsu 18-66
Record Dates: First submitted 2008-09-12; First posted 2008-09-15 (Estimated); Last update posted 2011-09-07 (Estimated); Status verified 2009-04

CONDITIONS: Non-small Cell Lung Cancer
Keywords: non-small cell lung cancer; previously untreated
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Sildenafil Citrate; Paclitaxel; Carboplatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Active Comparator): Sildenafil plus carboplatin and weekly paclitaxel
  Interventions: Drug: sildenafil; Drug: paclitaxel (taxol); Drug: carboplatin (palaplatin)
- P (Placebo Comparator): carboplatin and weekly paclitaxel
  Interventions: Drug: placebo; Drug: paclitaxel (taxol); Drug: carboplatin (palaplatin)

INTERVENTIONS:
Drug: sildenafil — 50mg, day1,8 and 15 in each cycle
  Arms: A
Drug: placebo — 1 tab, day 1,8 and 15 in each cycle.
  Arms: P
Drug: paclitaxel (taxol) — paclitaxel; 70mg/m2 div on day 1, 8 and 15, every 28 days
  Other Names: taxol
Drug: carboplatin (palaplatin) — carboplatin; AUC=6 on day 1, every 28 days
  Other Names: palaplatin

SUMMARY:
A comparison of combination chemotherapy of sildenafil plus carboplatin and weekly taxol with carboplatin and weekly taxol in patients with previously untreated advanced non-small cell lung cancer. The study hypothesis is that sildenafil may improve the distribution and efficacy of cytotoxic anticancer agents.

DETAILED DESCRIPTION:
Sildenafil is one of selective phosphodiesterase type 5 inhibitors. It is used to block the degradative action of phosphodiesterase type 5 on cyclic GMP in the smooth muscle cells lining the blood vessels, which leads to smooth muscle relaxation in blood vessels and increases blood flow. Because phosphodiesterase type 5 is also present in the arterial wall smooth muscle within the lungs, phosphodiesterase type 5 inhibitors is also used for the treatment of pulmonary hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of histologically confirmed stage IIIB or IV non-small cell lung cancer
* Good performance status (ECOG 0-1)
* No previous treatment
* Adequate bone marrow, liver and renal functions
* Must be able to swallow tablets
* Provided written informed consent

Exclusion Criteria:

* Severe complications or a concomitant malignancy
* Contraindicated sildenafil, carboplatin or taxol
* Inappropriate patients for entry to this study, judged by the physicians

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2007-02; Primary Completion 2009-03 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
progression free survival | three-year

SECONDARY OUTCOMES:
overall response rate | three-year

CONTACTS AND LOCATIONS:
Overall Officials: Kingo Chida, MD,PhD, Study Chair — Hamamatsu University School of Medicien Institution Review Board
Locations (1):
- Hamamatsu University School of Medicine, Hamamatsu, Japan